CLINICAL TRIAL: NCT07076589
Title: A Comparative Study Between the Usage of Flexible and Navigable Suction Ureteral Access Sheath (FANS) Versus Traditional Access Sheath in RIRS : Randomized Controlled Trial
Brief Title: A Comparative Study Between the Usage of Flexible and Navigable Suction Ureteral Access Sheath Versus Traditional Access Sheath in Retrograde Intrarenal Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yosseif elhousseiny ammar ahmed (Other)
Responsible Party: Sponsor-Investigator, Yosseif elhousseiny ammar ahmed, Principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-210-2025
Record Dates: First submitted 2025-06-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Stones, Kidney; Ureter Stones
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Using FANS (Active Comparator): After the successful induction of anesthesia, the lithotomy position will be adopted. Ureteroscopy will be used with the aid of a safety guidewire to evaluate the condition of the ureter. The serial dilation of the ureter using ureteral dilators up to 14 Fr . The FANS will be then inserted into the ureter under the guidance of the safety guidewire. The FANS tip will be positioned in the renal pelvis or calyces near the location of the stone.
  The FANS will be connected to a vacuum device, and the negative pressure will be applied. The actual intraoperative negative pressure value will be adjusted by the urologist through a pressure adjustment vent as needed. The irrigation volume was set using peristaltic pumps. Lithotripsy will be conducted using the holmium: yttrium aluminum garnet laser applying the dusting technique of laser lithotripsy. During lithotripsy, the FANS will allow us to retrieve most of the fragmented stone particles by application of the suction pressure. All cases w
  Interventions: Procedure: FURS
- Using traditional UAS (Active Comparator): The method of anesthesia, patient positioning, ureteral dilation, and lithotripsy were the same as those used in the FANS group.
  For the traditional UAS group, the end of the UAS will be positioned underneath the ureteropelvic junction (UPJ). The irrigation volume is applied using peristaltic pumps. The dusting technique of laser lithotripsy will be applied to the stones.
  All cases will be stented using JJ stents with the suitable size.
  Interventions: Procedure: FURS

INTERVENTIONS:
Procedure: FURS — FURS using traditional UAS & FANS

SUMMARY:
A comparative study between the Usage of Flexible and Navigable Suction Ureteral Access Sheath (FANS) versus Traditional Access sheath in RIRS : Randomized controlled trial .

DETAILED DESCRIPTION:
Urinary calculus is a worldwide urological disease, with a prevalence ranging from 1% to 13% in different regions . Currently, the main therapeutic methods beyond conservative treatment for renal calculi include extracorporeal shock wave lithotripsy (ESWL) and minimally invasive endoscopic surgical methods, including percutaneous nephrolithotomy (PCNL) and retrograde intrarenal surgery (RIRS). Treatment plans depend on the characteristics of calculi, patient factors, surgeon experience and the condition of medical centers .

Technological advancements in RIRS have been numerous in recent years, with the introduction of single-use flexible ureteroscopes and higher-power lasers being the most notable. High intrarenal pressure (IRP) can lead to pyelovenous backflow and infection from transient bacteraemia, particularly during laser lithotripsy. Another major concern is the retention of residual fragments (RFs), which are pieces that are hidden from view because of the snow-globe effect .

Therefore, in order to facilitate the clearance of RF and enhance the overall performance of RIRS, a variety of adjuncts have been developed, including pressure sensors to regulate IRP, a direct in-scope vacuum technique to aspirate dust, and stone retrieval devices that utilize suction technologies .

These objectives are all designed to achieve the triumvirate of successful RIRS: a high stone-free rate (SFR), minimal ancillary interventions, and minimal complications-the ultimate goal of all RIRS surgeons .

The ureteral access sheath (UAS) has been used in RIRS to reduce IRP and hence infectious complications, as well as to improve drainage, stone clearance, and intraoperative vision, thus shortening operative time. However, there still remains some debate over the ideal UAS size - too large risks injuring the ureteral mucosa and causing ischaemia, while too small defeats its purpose of improving drainage .

The addition of suction to a traditional UAS resulted in the conception of suction ureteral access sheath (SUAS). As demonstrated in clinical studies, the SUAS has the potential to reduce intrarenal temperature and pressure, thus reducing infectious complications and improving SFR .

Nevertheless, the SUAS continues to exhibit certain constraints . If it is positioned below the uretero-pelvic junction (UPJ), as is the case with the traditional UAS, the application of suction results in the collapse of the proximal ureteral mucosa. This reduces the calibre of the narrow UPJ and impedes the aspiration of RF by acting as a functional valve to block the opening of the UAS. Despite being positioned across the UPJ, it is incapable of overcoming acute angles or reaching distant calyces to facilitate the complete aspiration of particulate that has settled in dependent calyces .

A flexible-tip SUAS, also known as the flexible and navigable suction UAS (FANS), was developed as a natural evolution. This SUAS could be navigated using the flexible scope. FANS can be securely maneuvered into individual calyces under fluoroscopic guidance to remove fragments and dust more thoroughly and targeted through suctioning .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥14 years old in patients not known to have stone forming medical conditions.
* Renal stones diameter of ≤2 cm confirmed by CT with all types of configurations (branching & non-branching).
* Non - recurrent cases with no history of previous open renal surgeries or PCNL with normal renal anatomy.
* Patients with non - infected urine analysis.

Exclusion Criteria:

* Patients with abnormal urinary tract anatomy (such as horseshoe kidney or ileal conduit).
* Patients with medical conditions promoting stone formation (hyperparathyroidism - gout).
* Patients with history of stones on the same side with previous open surgical intervention or PCNL .
* Patients with e-GFR < 60 ml / min.
* Patients with uncontrolled urinary tract infection.
* Patients with health or other factors that are absolute contraindications to RIRS.
* Patients who are unable to understand or complete trial documentation.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
• Stone-free rate (SFR). | 12 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Yehia Abdelaziz Mohammed, Professor of urology, Principal Investigator — Cairo University
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After finishing the study and for 1 whole year

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT07076589/Prot_SAP_000.pdf